CLINICAL TRIAL: NCT06440408
Title: Calculating Wall Shear Stress in Pulmonary Veins of Infants Using Cardiac Magnetic Resonance Imaging: A Pilot Study
Brief Title: Calculating Wall Shear Stress in Infant Pulmonary Veins
Acronym: PVS-WSS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Ryan Callahan, MD, Assistant Professor of Pediatrics, Children's Hospital of Philadelphia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB 23-021612
Record Dates: First submitted 2024-05-24; First posted 2024-06-03 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary Vein Stenosis
Keywords: Cardiac Magnetic Resonance Imaging; Wall Shear Stress
MeSH Terms: conditions — Stenosis, Pulmonary Vein | interventions — Ferrosoferric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ferumoxytol enhanced cMRI (Experimental): A one time dose of Ferumoxytol will be administered prior to the cMRI in order to enhance the images. A dose of 4 mg/kg (max dose 510 mg) administered at a concentration of 8 mg/mL (in saline) will be used for this study. If the volume being administered is less than 6 mL, this is diluted with 3 mL of normal saline prior to administration. The drug is given over 15 minutes intravenously through a central or peripheral line. The drug is given at least 15 minutes prior to cardiac imaging.
  Interventions: Drug: Ferumoxytol

INTERVENTIONS:
Drug: Ferumoxytol — Ferumoxytol will be used as a contrast agent for the cMRI
  Other Names: Feraheme

SUMMARY:
The purpose of this study is to better understand pediatric pulmonary vein stenosis (PVS), which is the narrowing of blood vessels that connect the lungs to the heart. PVS is a life-threatening disease without a clear cause. The investigators think patients who develop PVS have an increased Wall Shear Stress (WSS) level in the pulmonary veins, which is the force placed on the walls of the veins. This study will determine if WSS can be calculated in the pulmonary veins of infants using Ferumoxytol enhanced Cardiac Magnetic Resonance Imaging (FcMRI). If possible, the investigators aim to use FcMRI to better screen patients at risk of PVS and to help guide therapy in patients with PVS.

DETAILED DESCRIPTION:
Background:

The mechanism of pediatric intraluminal pulmonary vein stenosis (PVS) remains unknown. It is hypothesized that elevated wall shear stress (WSS) as a result of excessive pulmonary blood flow (left to right shunts) and/or pulmonary vein distortion from surrounding anatomy contributes to the neo-intimal proliferation. Calculating WSS in pediatric pulmonary veins using ferumoxytol enhanced cardiac magnetic resonance (FcMRI) has not been reported and would represent a novel method of evaluation.

Objectives:

The primary objective is to determine the feasibility of calculating WSS in infant pulmonary veins using FcMRI. The secondary objective is to determine the magnitude and variability of WSS in pulmonary veins among high-risk patients and normal controls.

Study Design:

Prospective, interventional, single center, feasibility study

Setting/Participants:

Single center study at The Children's Hospital of Philadelphia. High-risk infants (n = 10) will include two groups of patients; (1) infants with moderate to severe bronchopulmonary dysplasia (BPD) and (2) infants with postoperative repair of total anomalous pulmonary venous connection (TAPVC). Group 1 participants will be infants who are undergoing an MRI as part of clinical care for other issues (i.e., MRI brain for hypoxic ischemia encephalopathy), with the research FcMRI being performed following the clinical care MRI. Group 2 participants will be infants who are undergoing FcMRI as part of clinical care. Controls (n = 10) will be pediatric patients without intracardiac defects who are undergoing FcMRI as part of clinical care (i.e., evaluation of anomalous coronary, aortopathy, vascular ring).

Study Procedures, Interventions and Measures:

Participants will undergo FcMRI and have the WSS calculated in each pulmonary vein (right upper, right lower, left upper, left lower) using several methodologies. Patients will be followed for 12 months following cMRI monitoring for a new diagnosis of PVS.

ELIGIBILITY:
Normal (Controls) Subjects Inclusion Criteria

1. Males or Females less than 18 years of age.
2. Weight > 3 kg.
3. Undergoing cMRI with ferumoxytol as part of clinical care.
4. Structurally normal heart (by echocardiography) with exception of small left to right shunts, isolated valve pathology, anomalous coronary arteries, extracardiac vascular anomalies such as arch anomalies.
5. Parental/guardian permission (informed consent).

Normal (Controls) Subjects Exclusion Criteria

1. Congenital heart disease (except small left to right shunts, isolated valve pathology, anomalous coronary arteries, extracardiac vascular anomalies such as arch anomalies).
2. Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.
3. Patient not receiving ferumoxytol as part of their cMRI due to a known hypersensitivity to the drug, or a known diagnosis of iron overload.

High-Risk Subject Inclusion Criteria

1. Males or Females less than 12 months of age.
2. Diagnosis of moderate to severe BPD (group 1) or TAPVC s/p repair (group 2).
3. Weight > 3 kg.
4. Undergoing non-contrast MRI for clinical reasons (group 1) or undergoing cMRI with ferumoxytol as part of clinical care (group 2).
5. Parental/guardian permission (informed consent).

High-Risk Subject Exclusion Criteria

1. Congenital heart disease with single ventricle physiology.
2. Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.
3. Patient has a contraindication to ferumoxytol such as a known hypersensitivity to the drug, or a known diagnosis of iron overload.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Wall Shear Stress level in infant pulmonary veins using cMRI | 12 months
  WSS (dyn/cm2) will be reported in each pulmonary vein using multiple modalities with data from the cMRI. This includes computational fluid dynamics, 4D-Flow and 4*Mu*v/r, where Mu is the viscosity of blood, r is the vessel radius, and v is the average velocity of blood.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Callahan, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hammer PE, McEnaney K, Callahan R, Baird CW, Hoganson DM, Jenkins KJ. The Role of Elevated Wall Shear Stress in Progression of Pulmonary Vein Stenosis: Evidence from Two Case Studies. Children (Basel). 2021 Aug 25;8(9):729. doi: 10.3390/children8090729. PMID 34572161
- [Background] Misra S, Fu AA, Misra KD, Glockner JF, Mukhopadhyay D. Wall shear stress measurement using phase contrast magnetic resonance imaging with phase contrast magnetic resonance angiography in arteriovenous polytetrafluoroethylene grafts. Angiology. 2009 Aug-Sep;60(4):441-7. doi: 10.1177/0003319709335908. Epub 2009 Jul 21. PMID 19625275
- [Background] Kamada H, Nakamura M, Ota H, Higuchi S, Takase K. Blood flow analysis with computational fluid dynamics and 4D-flow MRI for vascular diseases. J Cardiol. 2022 Nov;80(5):386-396. doi: 10.1016/j.jjcc.2022.05.007. Epub 2022 Jun 17. PMID 35718672
- [Background] Callahan R, Gauvreau K, Marshall AC, Sena LM, Baird CW, Ireland CM, McEnaney K, Bjornlund EC, Mendonca JT, Jenkins KJ. Outcomes in Establishing Individual Vessel Patency for Pediatric Pulmonary Vein Stenosis. Children (Basel). 2021 Mar 10;8(3):210. doi: 10.3390/children8030210. PMID 33802089
- [Background] Nguyen KL, Yoshida T, Kathuria-Prakash N, Zaki IH, Varallyay CG, Semple SI, Saouaf R, Rigsby CK, Stoumpos S, Whitehead KK, Griffin LM, Saloner D, Hope MD, Prince MR, Fogel MA, Schiebler ML, Roditi GH, Radjenovic A, Newby DE, Neuwelt EA, Bashir MR, Hu P, Finn JP. Multicenter Safety and Practice for Off-Label Diagnostic Use of Ferumoxytol in MRI. Radiology. 2019 Dec;293(3):554-564. doi: 10.1148/radiol.2019190477. Epub 2019 Oct 22. PMID 31638489